CLINICAL TRIAL: NCT02907775
Title: Multi-channel Stimulation for Post Stroke Spasticity (MUSTS): A Randomised Controlled Cross Over Feasibility Trial
Brief Title: Multi-channel Stimulation for Post Stroke Spasticity (MUSTS)
Acronym: MUSTS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sheffield Teaching Hospitals NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: STH19263
Record Dates: First submitted 2016-09-13; First posted 2016-09-20 (Estimated); Last update posted 2019-07-18 (Actual); Status verified 2019-07

CONDITIONS: Muscle Spasticity; Stroke
MeSH Terms: conditions — Muscle Spasticity; Stroke | interventions — Electrodes

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Transcutaneous Electric Nerve Stimulus (Active Comparator): Researcher 1 who is blind to patients' allocation group will perform the baseline assessments. The researcher 2 will determine the maximum tolerable level of stimulation. The researcher 2 will demonstrate to the participant how to apply the stimulation and will instruct the participant. The participant will revive the first intervention in the Royal Hallamshire Hospital under supervision of researcher 2. The researcher 2 will then issue the participants in Group-2 (SBS) with Shefstim and six multichannel electrodes. They will instruct each participant to change the electrode once every 3 days. On the 15th day the researcher 2 will visit them at home and issue further 6 multichannel electrodes and collect back the previous set. At the end of week 4, the patient will come to Hospital.
  Interventions: Device: Electrodes
- Sensory Barrage Stimulation (Active Comparator): Researcher 1 who is blind to patients' allocation group will perform the baseline assessments. The researcher 2 will determine the maximum tolerable level of stimulation. The researcher 2 will demonstrate to the participant how to apply the stimulation and will instruct the participant. The participant will revive the first intervention in the Royal Hallamshire Hospital under supervision of researcher 2. The researcher 2 will then issue the participants in Group-2 (SBS) with Shefstim and six multichannel electrodes. They will instruct each participant to change the electrode once every 3 days. On the 15th day the researcher 2 will visit them at home and issue further 6 multichannel electrodes and collect back the previous set. At the end of week 4, the patient will come to Hospital.
  Interventions: Device: ShefStim

INTERVENTIONS:
Device: ShefStim — Electrode arrays will be worn over the affected arm with stimulation applied over the extensor aspect of the upper arm
  Arms: Sensory Barrage Stimulation
Device: Electrodes — electrodes placed over the radial nerve in radial grove
  Arms: Transcutaneous Electric Nerve Stimulus

SUMMARY:
Over 87,000 people have a first stroke in the UK each year; about 70% of victims have altered arm function and about 40% are left with a non-functional arm. Spasticity is a significant deterrent for recovery of arm function following stroke. One in four patients develop spasticity within the first 2 weeks of the stroke and by 12 months 39 % have spasticity. The use of oral antispasticity medications like baclofen and tizanidine are often restricted due to side effects like sedation, weakness and floppiness. Compliance of adults to treatment with oral anti spasticity drugs is only around 50%.

There are a few exploratory studies on sensory stimulation using Transcutaneous Electrical Nerve Stimulation (TENS) in reducing spasticity. Amatya et al reviewed the evidence and concluded that there was not sufficient evidence to recommend its routine use. One possible explanation for the ineffectiveness of TENS is that it uses a single channel, single strength and fixed duration stimulation to which the nervous system may get habituated. We have developed Shefstim; a unique miniaturised 64 channel electrical stimulator. Using Shefstim we pioneered a technique called Sensory Barrage Stimulation ;rapid simultaneous stimulation at multiple sites, in a constantly changing pattern. We hypothesise that this approach will significantly reduce habituation compared to single site stimulation, thus providing a better treatment for spasticity.

Objective of the proposed study is to to explore the feasibility of conducting a community based randomised cross over trial comparing SBS with TENS for post stroke upper limb the spasticity of elbow flexors to optimise the stimulation parameters through quantifying objectively the muscular response to two different stimulation protocols.

DETAILED DESCRIPTION:
We will assess the safety and feasibility of delivering SBS and TENS for upper limb spasticity in the community. The trial is considered single blind as the assessor will be blinded as to the intervention. The investigator delivering the intervention cannot be blinded but will not be involved in the assessment of outcomes.

Twenty men and women will be randomised to receive either SBS or TENS. Participants will be identified from the stroke clinics, Community physiotherapy services, Assessment and Rehabilitation Centre and Functional Electrical Stimulation clinic in Sheffield. The treating team will identify the potential participants and will give them the information leaflet about the study. A member of the study team will then contact the participants between 7 and 14 days. Those who agree to participate in the study will be invited to attend a face to face appointment with a member of the study team at Royal Hallamshire Hospital.

Visit-1: During this visit the participant will be given opportunity to discuss the study and any concerns regarding the trial with the principal investigator. After this principal investigator will obtain the informed consent.

The participant will be asked to perform Action Research Arm test ( ARAT) which include a set of activities like grasping, holding and lifting objects with both affected and unaffected arms while we record the activity of 16 arm muscles using electromyography and motion sensors. This involves sticking small sensors on various muscles. The participant will then receive two different paradigms of SBS for 10 minutes each with a gap of 10 minutes in between and the effect on EMG will be recorded. The participant or carer will be trained to record the severity of spasticity in a diary between 6pm and 9pm on a scale ranging from 0 to 10; 0- no spasticity, 10 worst spasticity you can imagine.

Visit-2: The participant will be randomly allocated to either group-1 or group-2 using an online randomisation system. A researcher is blind to the allocation will do the assessments. Another researcher will deliver the intervention. Participants in group-1 will receive TENS and those in group-2 will revive SBS over extensor aspect of upper arm for one hour. The strength for stimulation will be just below the motor threshold or the maximum tolerable stimulation which ever is lower. The stimulation can cause a tingling sensation. Some people may find these stimulations slightly unpleasant. The researcher will again assess and will also look for any adverse event after the intervention. Participant or carer will be trained to apply the electrodes and deliver the intervention for 1 hour a day for next 4 weeks.

Visit 3: The researcher will again assess the participants and will also look for any adverse event after the intervention. Participant\carer will be asked to continue to record the severity of spasticity in a diary for next one week.

Visit-4: After assessment the participants in group-1 will receive TENS and in group-2 will receive SBS for one hour. As during the visit 2, the blinded researcher will check for any adverse events and assess the outcome measures after the stimulation. The participant or carer will be trained to apply the electrodes and deliver the intervention for 1 hour a day for next 4 weeks.

Visit 5: The blinded researcher will again assess the outcome measures and will also look for any adverse event after the intervention.

Interventions: This will occur in three phases.

Phase 1: Subjects will randomly be allocated to Group-1 to receive TENS, or Group-2 to receive SBS, for 60 minutes each day for four weeks. We will use a remote randomisation through telephone.

Researcher-1 who is blind to patients' allocation group will perform the baseline assessments. The researcher -2 will determine the maximum tolerable level of stimulation. The researcher-2 will demonstrate to the participant and \or the carer how to apply the stimulation and will instruct the participant. The participant will revive the first intervention in the Royal Hallamshire Hospital under supervision of researcher-2. The researcher-2 will then issue the participants in Group-2 ( SBS) with Shefstim and six multichannel electrodes. He \she will instruct each participant to change the electrode once every 3 days. On the 15th day the researcher-2 will visit them at home and issue further 6 multichannel electrodes and collect back the previous set. At the end of week 4, the patient will come to Royal Hallamshire Hospital.

The researcher-2 will collect all the electrodes and the equipment back. The researcher-1 will do all the outcome assessments.

Phase 2: No intervention period of two weeks.

Phase 3: Group-1 to receive SBS, or Group-2 to receive TENS, for 60 minutes each day for four weeks.

The first session of SBS and TENS will take place in Royal Hallamshire Hospital.

SBS group: We will use the stimulation techniques tested out in our previous study. Electrode arrays will be worn over the affected arm with stimulation applied over the extensor aspect of the upper arm. At the start of first session, stimulation will be increased over the arrays until movement is first observed. The stimulation level will then be set at 90% of this value, or the maximum tolerable if pain is reported and the value recorded. Stimulation will continue at this level moving around the array electrodes with a pseudo-random pattern for 60 minutes daily for 4 weeks. TENS group: We will use the stimulation techniques tested out in the previous studies, including our trial. Two surface electrodes will be placed over the radial nerve in radial grove. The intensity of stimulation will be set to 90% of the motor threshold. TENS will be applied for 60 minutes daily for 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 and above;
* Six months after stroke;
* Spasticity at elbow of grade-2 or more on the modified Ashworth scale.

Exclusion Criteria:

* Cognitive impairment that would interfere with their ability to comply with the experimental protocol or provide informed consent;
* Dermatological, rheumatologic or orthopaedic illnesses of the affected arm interfering with movement of the elbow;
* Pre-existing severe systemic disorders like cardiovascular disease; active cancer or renal disease; end stage pulmonary or cardiovascular disease; psychiatric illness including severe alcohol or drug abuse and depression;
* Inability to perform the baseline assessments;
* Severe tactile hypersensitivity;
* Participation in other, spasticity related studies;
* Within 12 weeks of receiving Botulinum toxin injections;
* Uncontrolled epilepsy;
* Pace maker or any other implanted devices;
* Pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2016-09-30 (Actual); Primary Completion 2018-09-30 (Actual); Study Completion 2018-09-30 (Actual)

PRIMARY OUTCOMES:
upper limb function after four weeks of intervention measured by the Action Research Arm Test | 4 weeks

SECONDARY OUTCOMES:
muscle activity as measured using EMG | 4 weeks
measures of muscle tone | 4 weeks
  Modified Ashworth Scale
strength | 4 weeks
  Medical Research Council grading
impact of spasticity | 4 weeks
  Leeds Arm Spasticity Scale-reference

CONTACTS AND LOCATIONS:
Overall Officials: Siva Nair, Principal Investigator — Sheffield Teaching Hospitals NHS FT
Locations (1):
- Sheffield Teaching Hospitals NHS FT, Sheffield, United Kingdom

IPD SHARING:
Plan to Share IPD: No